CLINICAL TRIAL: NCT06234956
Title: Open-label, Multi-centre, Non-Inferiority Study of Safety and Immunogenicity of BIMERVAX as Heterologous Booster for the Prevention of Coronavirus Disease 2019 (COVID-19) in Adolescents From 12 Years to Less Than 18 Years of Age.
Brief Title: Open-label, Multi-centre, Non-Inferiority Study of Safety and Immunogenicity of BIMERVAX for the Prevention of COVID-19 in Adolescents From 12 Years to Less Than 18 Years of Age.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hipra Scientific, S.L.U (Industry)
Collaborators: Veristat, Inc. (Other); VHIR (Unknown); Asphalion (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HIPRA-HH-3
Record Dates: First submitted 2023-10-20; First posted 2024-01-31 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BIMERVAX (Experimental)
  Interventions: Biological: BIMERVAX

INTERVENTIONS:
Biological: BIMERVAX — BIMERVAX

SUMMARY:
This is a Phase IIb, open-label, uncontrolled, multi-centre, non-inferiority clinical trial, to assess the safety and immunogenicity of BIMERVAX® as a heterologous booster dose in adolescents.

In this study a total of 300 adolescents from 12 to less than 18 years will be enrolled and followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged from 12 to less than 18 years at Screening.
* Participant's parent(s)/legal guardian(s) willing and able to sign the informed consent and can comply with all study visits and procedures. A written assent will be required for all participants in the study. Note: Participants are expected to be available for the duration of the study and whose parent(s)/legal guardian can be contacted by telephone during study participation.
* Participant must have received two previous doses of Comirnaty, last dose being at least 6 months before screening.
* Participant has a body mass index at or above the third percentile according to local Child Growth Standards at Screening Visit.
* Healthy participants and participants with pre-existing, chronic and stable diseases (non-immunocompromised), if these are stable and well-controlled according to the investigator's judgment, are eligible for inclusion in the study. Note: Healthy participants are determined by medical history, physical examination, and clinical judgment of the investigator. Healthy participants with pre-existing stable diseases, are defined as diseases not requiring significant change in the therapy or hospitalisation for worsening disease during the 6 weeks before enrolment.
* Has a negative Rapid Antigen Test (RAT) at Day 0 before BIMERVAX® vaccine administration.
* Participants biologically able to have children may be enrolled in the study if the participant fulfils all the following criteria:
* Has a negative urine pregnancy test at Screening (Day 0), only for those participants who are biologically able to become pregnant.
* Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the booster dose, only for those participants who are biologically able to become pregnant.
* Has agreed to continue adequate contraception or abstinence through 3 months following the booster dose.

  1. Participants with female reproductive system:

     1. Hormonal contraception (progestogen only or combined: oral, injectable or transdermal (patch)
     2. Intrauterine device.
     3. Vasectomized partner (the vasectomized partner should be the sole partner for that participant).
     4. Condom.
  2. Participants with male reproductive system:

     1. Vasectomized participants.
     2. Agree to use a condom in partners biologically able to become pregnant.
* Participant must have a body weight >50 kg at Screening visit to be eligible for the cellular immunology assays.

Exclusion Criteria:

* Acute illness with fever ≥ 38.0°C at Screening or within 24 hours prior to vaccination. Participant can be rescheduled for Screening when they have completed 24 hours without fever. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator.
* Received medications intended to prevent or treat COVID-19 before Screening, except for Comirnaty vaccines.
* Previous or current diagnosis of MIS-C.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behaviour or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Note: This includes both conditions that may increase the risk associated with study intervention administration or a condition that may interfere with the interpretation of study results.

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g. anaphylaxis) to any component of the study intervention(s).
* Immunocompromised individuals defined as those with primary and secondary immune deficiencies and those receiving chemotherapy or immunosuppressant drugs other than steroids and glucocorticoids (maximum 1 mg/kg/day of prednisone or total dose of 20mg/day by any administration route for a maximum of 30 consecutive days), within 90 days prior to vaccination or during the study.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Female who is pregnant or breastfeeding.
* Receipt of blood/plasma products, immunoglobulin, monoclonal antibodies, or receipt of any passive antibody therapy, within 90 days prior to vaccination or during the study.
* Participation in other studies involving study intervention within 28 days prior to screening and/or during study participation.
* Received any non-study vaccine (including seasonal Influenza vaccine) within 14 days before or after screening. For live or attenuated vaccines, 4 weeks before or after screening.
* History of illegal substance use or alcohol abuse within the past 2 years.
* History of a diagnosis or other conditions that, in the judgment of the investigator, may affect study endpoint assessment or compromise participant safety.
* Individuals who are family members of the Investigators.
* Individuals with documented medical history of microbiologically confirmed COVID-19 will not be eligible for the immunogenicity group.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 242 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Changes in immunogenicity against Omicron BA.1 | 14 days
  Neutralisation titre against Omicron BA.1 measured as inhibitory concentration 50 (IC50) by PBNA and reported as log10 concentration for each individual sample at Baseline and Day 14.
Changes in immunogenicity against Omicron BA.1 | 14 days
  Geometric Mean Titre (GMT) for group comparison with HIPRA-HH-2 at Baseline and Day 14.
Incidence of solicited local and systemic reactions (Safety and tolerability of PHH-1V) | 7 days
  Solicited local and systemic reactions through Day 7 after vaccination.
Incidence of unsolicited local and systemic adverse events (Safety and tolerability of PHH-1V) | 28 days
  Unsolicited local and systemic adverse events (AEs) through Day 28 after vaccination.
Incidence of related adverse events and serious adverse events (Safety and tolerability of PHH-1V) | 1 year
  Related adverse events (AEs) and all serious adverse events (SAEs) through the end of the study.
Incidence of adverse events of special interest (Safety and tolerability of PHH-1V) | 1 year
  Adverse event of special interest (AESI) through the end of the study.
Incidence of related medically attended adverse events (Safety and tolerability of PHH-1V) | 1 year
  Related medically attended adverse events (MAAE) through the end of the study.
Incidence of Grade 2, Grade 3 and Grade 4 changes in safety laboratory parameters (Safety and tolerability of PHH-1V) | 14 days
  Grade 2, Grade 3 and Grade 4 changes from Baseline in safety laboratory parameters through Day 14 after vaccination.

SECONDARY OUTCOMES:
Changes in immunogenicity against VOCs | Days 14, 84, 168 and 336
  Neutralisation titre against VOCs (at least Beta and Delta) measured as IC50 by PBNA and reported as log10 concentration for each individual sample at Baseline and Days 14, 84, 168 and 336.
Changes in immunogenicity against VOCs | Days 14, 84, 168 and 336
  GMT at Baseline and Days 14, 84, 168 and 336.
Changes in immunogenicity against Omicron BA.1 and VOCs | Day 14
  GMFR in neutralising antibodies titres against Omicron BA.1 and VOCs (at least Beta and Delta) at Baseline and Day 14.

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital Vall Hebron, Barcelona, Barcelona
  - CAP Centelles, Centelles, Barcelona
  - Hospital Josep Trueta, Girona, Girona
  - CAP Peralada, Peralada, Girona
  - Hospial HM Montepríncipe, Boadilla del Monte, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital HM Puerta del Sur, Móstoles, Madrid

IPD SHARING:
Plan to Share IPD: No